CLINICAL TRIAL: NCT04026984
Title: Double Blind, Multi-center Study to Evaluate the Safety and Efficacy of 100 mg Twice Daily Rifamycin SV MMX® Added to Standard ORT Versus Placebo Plus ORT, in the Treatment of Traveler's Diarrhea in Children Age 6 to 11 Years
Brief Title: Evaluate Safety and Efficacy of Rifamycin SV MMX in the Treatment of Traveler's Diarrhea in Children Age 6 to 11 Years
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-01-11/29
Record Dates: First submitted 2019-07-12; First posted 2019-07-19 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Traveler's Diarrhea
MeSH Terms: interventions — rifamycin SV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifamycin SV MMX plus ORT (Experimental): One tablet contains 50 mg Rifamycin SV-MMX® plus standard of care Oral Rehydration Therapy (ORT). Two 50mg tablets will be administered twice daily.
  Interventions: Drug: Rifamycin SV-MMX
- Placebo tablets plus ORT (Placebo Comparator): Matching placebo tablets plus standard of care Oral Rehydration Therapy (ORT)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifamycin SV-MMX — 2 Rifamycin SV-MMX® 50 mg tablets b.i.d. plus ORT
  Other Names: Rifamycin
  Arms: Rifamycin SV MMX plus ORT
Drug: Placebo — Matching Placebo tablets
  Arms: Placebo tablets plus ORT

SUMMARY:
This will be a double-blind comparative study, performed in pediatric subjects (Age 6-11) traveling to developing regions with a known high incidence of traveler's diarrhea. The subjects will be suffering from acute diarrhea for at least 12 hours, without symptoms of systemic infection.

DETAILED DESCRIPTION:
Approximately 142 subjects are expected to be enrolled in the study, 1:1 in the Rifamycin SV MultiMatrix (MMX) plus Oral Rescue Therapy (ORT) group and in the placebo tablets plus ORT group respectively. The day of randomization (Visit 1, Day 1), the subjects will start the treatment receiving ORT plus Rifamycin SV MMX 100 mg (as two tablets of 50 mg each) twice daily (morning and evening) or ORT plus placebo tablets (as two tablets) twice daily (morning and evening). The subjects will begin the treatment within 72 hours of onset of diarrhea. Treatment duration will last 72 hours. The total number of tablets for the entire treatment course will be 12 (4 × 50 mg tablets/day for 3 days). The administration of the ORT will follow the specification reported in the product label. The tablets will be orally administered during the day. No tablet administration will be done during the night.

After enrollment, subjects/their parents/or guardians will complete Diary cards (PDC) in which will be daily recorded date, time of first tablets intake, time and consistency of each stool, presence of blood in stools, abdominal pain/cramps, flatulence, tenesmus, urgency, nausea, vomiting, fever, adverse events (AEs), and concomitant medications.

During the study, the subjects will be assessed for safety and efficacy at Visit 2 (Day 2) and Visit 3 (Day 4/5) as final Study Visit.

Stool samples for microbiological assessment will be collected at Visits 1 and 3. Stool will be examined and cultured at local labs for main enteropathogens and for the presence of protozoa, ova and yeasts.

Blood and urine sampling for routine safety analyses will be collected at Visit 1 and at Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute bacterial diarrhea defined as at least 3 unformed stools within the 24 hours preceding randomization, with a duration of illness ≤72 h. The bacterial origin of diarrhea will be confirmed "a posteriori" by stool microbiology sampling at the time of screening.
* Presence of one or more signs or symptoms of enteric infection, including nausea, vomiting, abdominal cramps or pain, tenesmus, urgency
* History of recent travel from an industrialized country to a developing region with a known high incidence of travelers' diarrhea
* Male or female 6-11 years of age, providing an unformed pre-treatment stool
* The parent or legally acceptable representative must provide informed consent for the subject. The Subject must also provide written informed assent and be accompanied by the parent or legal guardian at the time of assent/consent signing.

Exclusion Criteria:

* Fever (>100.4ºF or 38ºC), or presence of signs and symptoms of systemic infection
* Known or suspected infection with non-bacterial pathogen
* Symptoms of acute diarrhea of >72 hours duration
* Presence of grossly bloody stool
* Moderate to severe dehydration
* History of inflammatory bowel disease (IBD)
* Abdominal ileus
* Severe dehydration
* Greater than two doses of an antidiarrheal medication within 24 hours before randomization, or any symptomatic therapy within 2 hours before enrolment
* Receiving antimicrobial drug with expected activity against enteric bacterial pathogens within the week prior to enrolment
* Hypersensitivity to rifamycin-related antibiotics or to any excipient included in the study medications
* Subjects unable/unwilling to comply with study protocol
* Participation in a clinical trial within the last 30 days

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Cure | 120 hours
  Passage of two or fewer soft stools and no watery stools, no fever (> 100.4 ºF or 38 ºC), and no signs or symptoms of enteric infection (other than mild excess gas/flatulence) during a 24-hour interval in the 120-hour data collection period after the first dose of study drug or Passage of no stools or only formed stools and no fever during a 48-hour interval in the 120-hour data collection period after the first dose of study drug, with or without other signs or symptoms of enteric infection.

SECONDARY OUTCOMES:
Time to last unformed stool (TLUS) | 120 hours
  defined as the interval in hours between the first dose of study drug and the last unformed stool passed, after which clinical cure was declared. Subjects who meet the criteria for clinical cure immediately after the start of the study and prior to passing any unformed stools are defined as having a TLUS of 0 hours. Subjects who terminated the study early due treatment failure will have a censored TLUS of 120 hours.
Microbiological Cure | 120 hours
  The proportion of subjects with an identified pathogen at baseline with microbiological eradication in the post-treatment stool sample.
Treatment Failure | 120 hours
  Defined as either of the following: Worsening diarrhea and/or signs or symptoms of enteric infection or failure to improve 24 hours or more after the first dose of study drug that results in administration of rescue therapy and/or Not achieving Clinical Cure in the 120-hr data collection period after the first dose of study drug or use of antimicrobial prohibited concomitant medication. Occurrence of AEs.

CONTACTS AND LOCATIONS:
Overall Officials: June Almenoff, MD, PhD, Study Director — RedHill Biopharma, Inc.